CLINICAL TRIAL: NCT00003122
Title: Phase II Trial of Surgery as the Only Treatment for INSS Stage 2A & 2B Neuroblastoma
Brief Title: Surgery in Treating Patients With Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065880; SIOP-95-1; EU-96053
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-07

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Procedure: surgical procedure

SUMMARY:
RATIONALE: Surgery may be an effective treatment for neuroblastoma.

PURPOSE: This phase II trial is studying how well surgery works in treating patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety and efficacy of surgical treatment alone for stage II neuroblastoma without N-myc amplification (NMA).
* Describe predictive factors of relapse and survival for stages I and II neuroblastoma without NMA treated by surgery alone.

OUTLINE: Patients with localized resectable tumors undergo surgery. Postoperative evaluations are performed 30 days following surgery. Study patients with stage I (without N-myc amplification) tumors and trial patients with stage II tumors receive no further therapy.

Study patients (except stage I patients) receive surgery and/or chemotherapy according to other protocols as necessary for disease progression or relapse.

Patients are followed every 3 months for the first year, then every 4 and 6 months for the second and third year respectively, then yearly for 5 years.

PROJECTED ACCRUAL: This study will accrue 140 stage II patients for the trial portion at a rate of 40 per year over 3.5 years. At least 70 more patients will be accrued for the study portion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Trial: Histologically proven International Neuroblastoma Staging System (INSS) stage IIA and IIB neuroblastoma without amplification of the N-myc oncogene
* Study: Histologically proven neuroblastoma

  * Stage I
  * Stage II with amplified N-myc
  * Stage II without evaluation of N-myc
  * Stage II with symptomatic spinal cord compression
  * Stage III
* No metastases diagnosed within 1 month of study

PATIENT CHARACTERISTICS:

Age:

* 20 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No adjuvant chemotherapy planned

Endocrine therapy:

* Prior use of steroids allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 1994-12

PRIMARY OUTCOMES:
Safety and efficacy
Predictive factors of relapse and survival

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marie Michon, MD, Study Chair — Institut Curie
Locations (96):
- Austria (6):
  - Universitaet Kinderklinik, Graz
  - Innsbruck Universitaetsklinik, Innsbruck
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - LKH Leoben, Leoben
  - St. Johanns-Spital, Salzburg
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
- France (25):
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - CHU de Caen, Caen
  - CHR Clermont Ferrand, Hotel Dieu, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Hopital Saint Antoine Lille, Lille
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Hopital, Paris
  - Hopital Jean Bernard, Poitiers
  - Hopital Americain, Reims
  - Hopital Sud, Rennes
  - Hopital Charles Nicolle, Rouen
  - CHU Sainte-Etienne - Hopital Nord, Saint-Étienne-d'Orthe
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Regional de Purpan, Toulouse
  - C.H. Bastien de Clocheville, Tours
  - CHRU de Tours - Hopital Trousseau, Tours
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Italy (27):
  - Universita Degli Studi di Bari, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Spedali Civili di Brescia, Brescia
  - Ospedale Oncologico A. Businco, Cagliari
  - Policlinico Dell'Universita, Catania
  - Ospedale Galliera, Genoa
  - Istituto Giannina Gaslini, Genoa
  - Istituti Clinici di Perfezionamento, Milan
  - Fondazione Istituto Nazionale dei Tumori, Milan
  - Ospedale Niguarda Ca'Granda, Milan
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Ospedale S.S. Annunziata Napoli, Naples
  - Federico II University Medical School, Naples
  - Clinica Pediatrica I, Naplesi
  - Azienda Ospedaliera di Padova, Padua
  - Clinica Pediatrica Palermo, Palermo
  - Azienda Ospedaliera Di Parma, Parma
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Ospedale Silvestrini, Perugia
  - Ospedale Santa Chiara Pisa, Pisa
  - Azienda Policlinico Umberto Primo, Rome
  - Ospedale Bambino Gesu, Rome
  - Clinica Ars Medica, Rome
  - Istituto Clinica Medica, Sassari
  - University of Siena, Siena
  - Clinica Pediatrica Trieste, Trieste
  - Ospedale Infantile Regina Margherita, Turin
- Netherlands (2):
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
- Spain (14):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Carlos Haya De Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital General de Galicia, Santiago de Compostela
  - Hospital Universitario La Fe, Valencia
  - Complejo Hospitalario Xeral de Vigo, Vigo Pontevedra
  - Hospital Des Cruces, Vizcaya
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Hopital des Enfants, Geneva
  - Ostschweizer Kinderspital, Sankt Gallen
- United Kingdom (18):
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Great Ormond Street Hospital for Children, London, England
  - University College of London Hospitals, London, England
  - Christie Hospital, Manchester, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Llandough Hospital, Llandough, Wales